CLINICAL TRIAL: NCT04963387
Title: Effects of Whole Body Vibrations on Functional Independence on Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Collaborators: Riphah International University (Other)
Responsible Party: Principal Investigator, Esha Khan, Senior Lecturer, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIPHAH/RCRS/REC/00517
Record Dates: First submitted 2021-07-05; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Older Adults With Moderate Balance Risk
Keywords: Balance; Whole Body Vibration; Berg Balance Scale; Older Adults; Physiotherapy

STUDY DESIGN:
Intervention Model Description: Single center, parallel group randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole body vibration (Experimental): Balance and muscle strengthening exercises with whole-body vibration, strengthening exercise included straight leg raise with weights, and balance training including walking heel to toe for 20 steps vibration exposure was given in 1-minute bouts, with rest period of one to two minutes between bouts, with the exposure whole body vibration for about four minutes on every session. The duration of vibration exposure was preset with the automatic set time intervals in the vibration machine Prior to each vibration bout. When the predefined time was reached the machine automatically turned off . Based on previous researches the total exposure of four minutes per session interval was selected. In this study frequency of 30Hz (4 weeks), with 0.9 mm vertical displacement was used.
  Interventions: Other: Whole body vibration
- Balance and Strengthening exercise (Active Comparator): Balance and strengthening exercises includes straight leg raise with weights 10 reps. and tandem walk 20 steps 3 days in week for 4 weeks
  Interventions: Other: Balance and Strengthening exercise

INTERVENTIONS:
Other: Whole body vibration — Balance and muscle strengthening exercises with whole-body vibration, strengthening exercise included straight leg raise with weights, and balance training including walking heel to toe for 20 steps. In this study frequency of 30Hz (4 weeks), with 0.9 mm vertical displacement was used.
  Arms: Whole body vibration
Other: Balance and Strengthening exercise — Balance and strengthening exercises includes straight leg raise with weights 10 reps. and tandem walk 20 steps 3 days in week for 4 weeks
  Arms: Balance and Strengthening exercise

SUMMARY:
Functional limitation and balance deficits occur with aging in normal healthy individuals due to decline in muscle strength. Muscle strengthening exercises and balance training has shown improvement of functional status of elderly. And whole body vibrations along with strengthen and balance training has been suggested to reduce the effects of aging in balance and functional abilities. Aim of this study was to find out the additional effects of whole body vibration along with balance training in older adults. It was a Randomized Control Trial Study. Study setting was railway general hospital Rawalpindi. Inclusion Criteria was Age 50 to 70 years old people, with moderate fall risk (BBS Score 21-40), both genders with Controlled diabetes and HTN, 112 Subjects were randomly and equally allocated to experimental group(n=56) and control group(n=56) through toss and coin method. Participants in both groups were examined for balance abilities with the Berg Balance Scale, Functional Independence Scale, & Timed up and Go Test (TUG) before and after 4 weeks treatment protocol.

DETAILED DESCRIPTION:
This study was a Randomized control trial. Conducted in Railway General Hospital Rawalpindi from January 2019 to July 2019. 300 older adults were screened and 112 were selected on the basis of inclusion criteria. Subjects were randomly allocated to control and experimental group through toss and coin method, 56 being in each group. Control group subjects received balance and strengthening exercises 3 times in a week for 4 weeks. While experimental group participants received same balance and strengthening exercises with whole body vibration 3 times in a week for 4 weeks. Vibration exposure was given in 1-minute bouts, with rest period of one to two minutes between bouts, with the exposure whole body vibration for about four minutes on every session, Balance exercises included tandem walk 20 steps and single leg raise with weights 10 repetition.(8,9) Tools used in this study were Berg Balance scale a 14 item scale. The score of each item ranges from zero to four, zero being the last point and 4 being the highest point the total score for these 14 items were 56. If the score is between 41 to56 then it is considered normal if it is from 20 to 40 the risk of balance deficits are moderate but if the score comes below 19 then risk of fall enhances. Almost 10 to 15 minutes are required to perform this scale on an individual. Functional Independence Measure It consisted of eighteen item; for motor items score 13 and five for cogitation which includes communication and cognition, each of the value is scored on a 7-point scale. The third tool used in this study was Time Up and Go test asses the static and dynamic balance it requires the time taken by individual to raise from a chair walk three meters, turn around walk back and sit on the chair. Subjects in both groups were pre assessed using these three tools and after completion of four weeks subjects were reassessed and the difference of score was noted. Data of this study was analyzed by using SPSS software version 25.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 to 70 years
* With moderate fall risk (BBS Score 21-40)
* Both genders
* Controlled diabetes and hyper tension

Exclusion Criteria:

* Patient with any type of surgical intervention which may hinder assessment or treatment
* Patient with any cognitive dysfunction.
* Patients with neurological disease (i.e. stroke, vestibular cochlear issue)
* Patients with any behavioral problem
* Patient with ischemic heart disease, Tumors

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Berg Balance Scale score | Baseline and 4 week
  14 item scale was established for elder population to asses balance deficits in them. The score of each item ranges from zero to four, zero being the last point and 4 being the highest point the total score for these 14 items were 56.
Change from Baseline in Functional Independence Scale score | Baseline and 4 week
  It consist of eighteen item; for motor items score 13 and five for cogitation which includes communication and cognition, each of the value is scored on a 7-point scale
Change from Baseline in Timed Up and Go test | Baseline and 4 week
  Define fall threat and assess the improvement of balance, sit to stand and walking.

CONTACTS AND LOCATIONS:
Overall Officials: Esha Khan, Principal Investigator — University of Lahore
Locations (1):
- Rehabilitation Department of Pakistan Railway Hospital Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No